CLINICAL TRIAL: NCT06897397
Title: Determination of the Effect of Case Management-Based Electronic Fetal Monitoring Training Given to Midwifery Students on EFM Monitoring Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Doç. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBU-AYDINKARTAL-010
Record Dates: First submitted 2024-12-07; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-12

CONDITIONS: Determining the Effect of Case Management-Based Electronic Fetal Monitoring Training Given to Midwifery Students on EFM Monitoring Self-Efficacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (n:40) (Experimental): Students will be provided with information about the education plan flow chart, education plan content, and environment. 40 students assigned to the intervention group will be provided with information about EFM training based on the case method. Before the application, all groups will be provided with 4 hours of theoretical information about EFM interpretation via a power point presentation.
  Interventions: Other: Case Study
- Control group (n:40 (No Intervention): Control group students will receive 4 hours of theoretical training. The training will be held in the midwifery department lecture hall.

INTERVENTIONS:
Other: Case Study — Students will be provided with information about the education plan flow chart, education plan content, and environment. 40 students assigned to the intervention group will be provided with information about EFM training based on the case method. Before the application, all groups will be provided with 4 hours of theoretical information about EFM interpretation via a power point presentation.
  Arms: Intervention group (n:40)

SUMMARY:
This study was planned to examine the effects of case management-based electronic fetal monitoring (EFM) training on midwifery students' EFM monitoring self-efficacy.

The research population will consist of second-year students studying at the Department of Midwifery, Hamidiye Faculty of Health Sciences (HSBF), Health Sciences University (SBÜ) in the spring semester of the 2023-2024 academic year (N: 80).

In this semi-experimental pre-test and post-test design and control group study, in order to determine the sample size; the data were normally distributed, the standard deviation of the main mass was estimated as 1 and the effect size (effect size, difference) was estimated as 0.8. For the analysis to be conducted, it was calculated that the highest power value of the study would be 0.942182 if two independent n₁=40, n₂=40 samples were taken at a significance level of 5%. The G-power analysis result is given below.

The students who volunteer to participate in the study will be assigned to the intervention and control groups with the computer-aided simple random sampling method. Computer-aided randomization will be used in the study, and the number of cases will be entered through the program with the URL address https://www.randomizer.org and random assignment will be made to the intervention and control groups. The study will be conducted single-blind. Before the application, all groups will be given 4 hours of theoretical information about EFM interpretation with a power point presentation. After the information, the "Electronic Fetal Monitoring Self-Efficacy Scale" will be applied as a pre-test. After the training, all students will be applied the "Electronic Fetal Monitoring Self-Efficacy Scale".

ELIGIBILITY:
Inclusion Criteria:

* Being a volunteer to participate in the research.
* Being an active student in the 2nd year of the Department of Midwifery, Hamidiye Faculty of Health Sciences, University of Health Sciences.

Exclusion Criteria:

- Being a passive student in the 2nd year of the Department of Midwifery, Hamidiye Faculty of Health Sciences, University of Health Sciences.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | 10 minutes
  This form, created by researchers based on literature, includes questions about the participants' age, high school graduation, case-based education status, etc.
Electronic Fetal Monitoring Self-Efficacy Scale | 10 minutes
  It is a scale that can be applied to health professionals and students in the health field. It is a 4-point Likert-type scale with 32 items, each item ranging from "Very confident" to "Not confident". Each item includes direct expressions and is calculated as Very confident = 4 points, Confident = 3 points, Somewhat confident = 2 points and Not confident = 1 point. A general score is obtained from the sum of all items. A high score indicates that EFM monitoring self-efficacy is high. The lowest score to be obtained from the scale varies between 32 and 128. The scale does not have a cut-off score.

SECONDARY OUTCOMES:
Introductory Information Form | 10 minutes
  This form, created by researchers based on literature, includes questions about the participants' age, high school graduation, case-based education status, etc.
Electronic Fetal Monitoring Self-Efficacy Scale | 10 minutes
  It is a scale that can be applied to health professionals and students in the health field. It is a 4-point Likert-type scale with 32 items, each item ranging from "Very confident" to "Not confident". Each item includes direct expressions and is calculated as Very confident = 4 points, Confident = 3 points, Somewhat confident = 2 points and Not confident = 1 point. A general score is obtained from the sum of all items. A high score indicates that EFM monitoring self-efficacy is high. The lowest score to be obtained from the scale varies between 32 and 128. The scale does not have a cut-off score.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No